CLINICAL TRIAL: NCT06730087
Title: Extravascular Lung Water and Fluid Responsiveness in Critically Ill Patient
Brief Title: Cardiometry in Hypotensive and Pumonary Congestion
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud, lecturer assistant, Assiut University
Other Study IDs: cardiometry in critically ill
Record Dates: First submitted 2024-11-06; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Shock; Pulmonary Congestion
Keywords: cardiometry
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2 groups which will compare cardiometry with ultrasound: patients will be divided into two groups: Group 1 patients with blood pressure less than 90/60 to assess fluid responsiveness and group 2 patients with sonographic finding of increase extravascular lung water in the form of interstitial edema or pulmonary edema or by electrical cardiometry (increase thoracic fluid content).

SUMMARY:
Assessment of validity of electrical cardiometry (EC) to measure fluid responsiveness and extravascular lung water that is expressed in the form of (thoracic fluid content) .

DETAILED DESCRIPTION:
1. Study Setting:

   The study will be conducted in Assiut University Hospital, in respiratory intensive care unit.

   This study is a cross sectional design for Extravascular lung water and fluid responsiveness assessment in critically ill patient
2. Study subjects:

   1. Inclusion criteria:

      1. Patients who are 18 years old or more.
      2. patients will be divided into two groups: Group 1 patients with blood pressure less than 90/60 to assess fluid responsiveness and group 2 patients with sonographic finding of increase extravascular lung water in the form of interstitial edema or pulmonary edema or by electrical cardiometry (increase thoracic fluid content).
   2. Exclusion criteria:

      1. Patients less than 18 years old.
      2. Patients who refuse to participate in the study.
   3. Sample Size Calculation:

      Sample size was calculated using the Buderer's formula for sensitivity and specificity of diagnostic health studies described by Zaidi et. al. 1 For Electrical Cardiometry in the fluid responsiveness group, the following inputs were used: expected sensitivity of Electrical Cardiometry in fluid responsiveness = 81%, expected specificity = 90%, expected sensitivity for ultrasound = 90% (8,9) , desired precision = 10%, and confidence level = 90%. The calculated sample size was 50 cases.

      For Electrical Cardiometry in the congestion group, the inputs were: expected sensitivity of Electrical Cardiometry in congestion = 89%, expected specificity = 83%, expected sensitivity for ultrasound = 88% (10,11),desired precision = 10%, and confidence level = 90%. The calculated sample size was 30 cases.
      1. Zaidi, S. M. H., Waseem, H. F., Ansari, F. A., Irfan, M., Fahim, S., & Ahmad, M. (2016, March). Sample size estimation of diagnostic test studies in health sciences. In Proceedings of 14th International Conference on Statistical Sciences (Vol. 29, pp. 239-246).
3. Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):

Methods:

Electrocardiometry:

The method of electrical cardiometry requires the use of 4 ECG electrodes, 2 attached to the left side of the neck and 2 attached at the lower thorax. An electrical alternating current (AC) of constant amplitude is applied via the pair of outer electrodes toward the thorax and in particular the ascending and descending aorta. Current is directed toward the aorta because blood is the most conductive material in the thorax. The ratio of applied current and measured voltage equals the conductivity (or bioimpedance), which is recorded over time. The steep increase in conductivity seen beat to beat is attributed to the orientation of red blood cells. The time when the slope is most steep is directly related to the peak aortic blood acceleration (12).

ICON® Parameters Blood Flow SV/SI HR CO/CI Stroke Volume / Stroke Index Heart Rate Cardiac Output /Cardiac Index Vascular System SVR /SVRI Systemic Vascular Resistance/ SVR-Index based on input of MAP and CVP Contractility ICON™ VIC™ STR Index of Contractility Variation of Index of Contractility Systolic Time Ratio (PEP/LVET) CPI Cardiac Performance Index Fluid Status TFC Thoracic Fluid Content SVV Stroke Volume Variation FTC Corrected Flow Time Oxygen Status DO2 / DO2I Oxygen Delivery / DO2-Index based on input of Hemoglobin and SpO2

IVC distensibility index:

In mechanically ventilated patients, the IVC distensibility index is calculated using the formula: IVC distensibility index = [(maximum diameter on inspiration-minimum diameter on expiration)/minimum diameter on expiration] (9). fluid responsiveness if it is > 18% (13).

Chest Ultrasonography A zone was considered positive for pulmonary congestion if ≥3 B-lines were shown (14).

Action plan and outcomes

1. All patients' data regarding age, gender, sex and essential diagnosis will be taken.
2. Patients' vital signs especially blood pressure and heart rate and rhythm.
3. Hemoglobin level will be acquired for all patients.
4. In intubated patients with blood pressure less than 90/60 fluid will be given500 mL crystalloids according Stroke volume variation (SVV) and thoracic fluid index. Fluid responsiveness was defined as SVV >10% to 15% suggests that the patient is fluid responsiveness as indicates that stroke volume is sensitive to fluctuations in preload caused by the respiratory cycle. Comparing fluid responsiveness first measurement between SVV by electrocardiometry and IVC distensibility. Other parameters of electrocariometery will be documented.
5. In patients clinically suspected pulmonary edema will be evaluated by ultrasonography and by electrical cardiometry
6. CVP will be measured.
7. Incidence of mortality, duration of MV and duration of ICU stay will be acquired for patients.

(4) Research outcome measures:

a. Primary (main): electric cardiometry effectiveness in fluid management in critically ill patient b. Secondary (subsidiary):

(5)Data management and analysis (Details needed): Data collection: medical records Computer software IBM SPSS software version 22.0 (SPSS Inc.,Chicago,IL) Statistical tests Statistical tests Normality of data will be assessed using Shapiro walk test. Normally distributed data will be represented as mean ± SD,median9range0 and numbers(%),chi square test or fisher's exac test will be used in categorical data .independent t-test will be used to compare between parametric data,Mann-Whitney will be used to compare non parametric values in the studied groups.p-value<0.05 will be considered statistically significant.

(6)References (max. 15) and written in Vancouver style:

1. Marik P, Bellomo R. A rational approach to fluid therapy in sepsis. BJA: British Journal of Anaesthesia [Internet]. 2016 Mar 1 [cited 2024 Jul 29];116(3):339-49. Available from: https://dx.doi.org/10.1093/bja/aev349
2. Rehberg S, Enkhbaatar P, Traber DL. Arginine vasopressin in septic shock: supplement or substitute for norepinephrine? Crit Care. 2009;13(4):178.
3. Marik PE, Baram M, Vahid B. Does central venous pressure predict fluid responsiveness? A systematic review of the literature and the tale of seven mares. Chest [Internet]. 2008 [cited 2024 Jul 29];134(1):172-8. Available from: https://pubmed.ncbi.nlm.nih.gov/18628220/
4. Magder S. Fluid status and fluid responsiveness. Curr Opin Crit Care [Internet]. 2010 Aug [cited 2024 Jul 29];16(4):289-96. Available from: https://pubmed.ncbi.nlm.nih.gov/20543685/
5. Cherpanath TGV, Lagrand WK, Schultz MJ, Groeneveld ABJ. Cardiopulmonary interactions during mechanical ventilation in critically ill patients. Neth Heart J [Internet]. 2013 Apr [cited 2024 Jul 29];21(4):166-72. Available from: https://pubmed.ncbi.nlm.nih.gov/23460128/
6. Cherpanath TGV, Geerts BF, Lagrand WK, Schultz MJ, Groeneveld ABJ. Basic concepts of fluid responsiveness. Netherlands Heart Journal [Internet]. 2013 Dec [cited 2024 Jul 29];21(12):530. Available from: /pmc/articles/PMC3833913/
7. Summers RL, Shoemaker WC, Peacock WF, Ander DS, Coleman TG. Bench to bedside: electrophysiologic and clinical principles of noninvasive hemodynamic monitoring using impedance cardiography. Acad Emerg Med [Internet]. 2003 Jun 1 [cited 2024 Jul 30];10(6):669-80. Available from: https://pubmed.ncbi.nlm.nih.gov/12782531/
8. Yao B, Liu JY, Sun YB, Zhao YX, Li L Di. The value of the inferior vena cava area distensibility index and its diameter ratio for predicting fluid responsiveness in mechanically ventilated patients. Shock. 2019 Jul 1;52(1):37-42.
9. Sharkawy MS El, Abdelghany MS, Dabe AA El, Hafez AAA El. Validation of Electrical Cardiometry Measurements Compared to Transthoracic Echocardiography in Fluid Responsiveness in Sepsis. J Adv Med Med Res. 2022 Apr 26;10-20.
10. Maw AM, Hassanin A, Ho PM, McInnes MDF, Moss A, Juarez-Colunga E, et al. Diagnostic Accuracy of Point-of-Care Lung Ultrasonography and Chest Radiography in Adults With Symptoms Suggestive of Acute Decompensated Heart Failure: A Systematic Review and Meta-analysis. JAMA Netw Open [Internet]. 2019 Mar 1 [cited 2024 Sep 16];2(3):e190703. Available from: /pmc/articles/PMC6484641/
11. Mahmoud KH, Mokhtar MS, Soliman RA, Khaled MM. Non invasive adjustment of fluid status in critically ill patients on renal replacement therapy. Role of Electrical Cardiometry. The Egyptian Journal of Critical Care Medicine. 2016 Aug;4(2):57-65.
12. ICON® - Portable Noninvasive Cardiometer │ OSYPKA MEDICAL [Internet]. [cited 2024 Aug 6]. Available from: https://www.osypkamed.com/products/electrical-cardiometry/icon/
13. Lujan Varas J, Martinez Díaz C, Blancas R, Martinez Gonzalez O, Llorente Ruiz B, Molina Montero R, et al. Inferior vena cava distensibility index predicting fluid responsiveness in ventilated patients. Intensive Care Medicine Experimental . 2015;3.
14. Dávila-Román VG, Checkley W. Lung Ultrasound in Cardiac Intensive Care. Circ Cardiovasc Imaging [Internet]. 2020 Jun 1 [cited 2024 Sep 4];13(6):E010909. Available from: https://www.ahajournals.org/doi/10.1161/CIRCIMAGING.120.010909

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years old or more.
2. patients will be divided into two groups: Group 1 patients with blood pressure less than 90/60 to assess fluid responsiveness and group 2 patients with sonographic finding of increase extravascular lung water in the form of interstitial edema or pulmonary edema or by electrical cardiometry (increase thoracic fluid content).

Exclusion Criteria:

1. Patients less than 18 years old.
2. Patients who refuse to participate in the study.

eria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in Assiut University Hospital, in respiratory intensive care unit.
  This study is a cross sectional design for Extravascular lung water and fluid responsiveness assessment in critically ill patient
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
electric cardiometry effectiveness in fluid management in critically ill patient | baseline
  compairing fluid responsiveness by stroke vloume variation in carddiometry( Fluid responsiveness was defined as SVV >10% to 15%) and IVC destinsability index by ultrasound (fluid rspnisveness was defined as [(maximum IVC diameter on inspiration-minimum diameter on expiration)/minimum diameter on expiration] > 18%). compairing pulmonary edema by fluid thoracic content(normal range:25 to 35) in cardiometry and B lines in chest ultrasound(more than 3 b-lines in all 4 fields/BLUE points considered positive for pulmonary edema according to BLUE protocol).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - faculty of mdicine Assiut university, Asyut, Asyut Governorate
  - faculty of medicine Assiut university, Asyut

IPD SHARING:
Plan to Share IPD: Undecided